CLINICAL TRIAL: NCT04641182
Title: Observational Study of Prone Position for Nonintubated Patients With COVID-19 and Hypoxemic Respiratory Failure
Brief Title: Prone Position for Nonintubated Patients With COVID-19 and Hypoxemic Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2020-09-12; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Ards; Respiratory Failure
MeSH Terms: conditions — COVID-19; Acute Lung Injury; Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prone position: Prone position per institutional protocol and as indicated by the treating physician
  Interventions: Other: Prone position
- No prone position: The control group will not be in prone position

INTERVENTIONS:
Other: Prone position — Prone position as indicated by the treating physician as specified in the institutional protocol
  Groups: Prone position

SUMMARY:
The aim of this observational study is to evaluate the physiological and clinical effects of prone position in awake patients with respiratory failure due to COVID-19.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the role of prone positioning in SARS-CoV-2 infected patients that are not intubated. Prone patient placement during invasive mechanical ventilation is a widespread practice in the management of severe ARDS. However, few attempts have been made to implement the prone position in patients that spontaneously ventilate with supplemental oxygen. Considering that it is a procedure that does not require additional equipment and does not represent an additional cost for its implementation, it becomes a valuable tool in the context of COVID-19 where intubation is associated with high mortality. The investigators will analyze a cohort of patients with COVID-19 and respiratory failure managed with prone position as indicated by the attending physician and register physiological variables and clinical outcomes (intubation and death).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with confirmed or suspected COVID-19 pneumonia requiring more than 3 liters per minute of supplemental oxygen or a Fraction of Inspired Oxygen (FIO2) over 35% to keep Pulse Oximetry Saturation (SpO2) over 90%
* Treating physician indicated prone position as instructed by the institutional protocol
* Patient capable of changing position with minimal help from the personnel

Exclusion Criteria:

* Patient requiring immediate intubation
* Patient requiring non-invasive mechanical ventilation
* Respiratory Rate > 40, signs of respiratory fatigue or unconsciousness with inability to protect the airway
* PaCO2 > 50mmHg
* Hemodynamic instability (defined by Heart Rate > 120, Systolic Pressure < 90mmHg, Mean Arterial Pressure < 60mmHg or requiring vasopressor support)
* Obesity with BMI > 40 (Body Mass Index: weight in kilograms and height in meters will be combined to attain BMI in kg/m2)
* Persistent vomiting
* Facial or thoracic trauma or recent surgery contraindicating the prone position
* Pregnancy > 20 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized COVID-19 adult patients with acute respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Therapeutic failure | At 14 days
  Defined by death or intubation or use of non-invasive ventilation
Mortality | At day 28
  Number of patients that die
Length of hospital stay | At 28 days
  Number of days spent by the patients at the hospital
Days requiring high flow nasal oxygen | At 28 days
  Number of days the patients require high flow nasal oxygen therapy
Days requiring supplemental oxygen | At 28 days
  Number of days the patients require supplementary oxygen
Displacement of invasive devices during position changes | At 28 days
  Unintentional displacement or removal of Invasive devices including : central and peripheric vascular catheters, urinary catheter and chest tubes
Occurrence of pressure ulcers on the anterior surface of the body | At 28 days
  Number of patients that develope pressure ulcers on the anterior surface of the body

SECONDARY OUTCOMES:
Respiratory superinfection | At 28 days
  Certified by a respiratory tract sample and culture
Delirium | At 28 days
  Defined by the Confusion Assessment Method (CAM)
Caloric intake | At 28 days
  Daily number of ingested calories (in kilocalories) by the patients is recorded
Proteic intake | At 28 days
  Daily number of ingested proteins (in grams) by the patients is recorded

OTHER OUTCOMES:
Dyspnea | At 28 days
  Using a scale from 1 to 10 (from 1 no dyspnea to 10 maximum dyspnea)
Comfort with the position | At 28 days
  Using a scale from 1 to 4 (1 is very comfortable and 4 is very uncomfortable)
Oxygen saturation | At 28 days
  Using PAFI (PAFI: Index calculated by Pressure of Arterial Oxygen / Inspired Fraction of Oxygen)
Oxygen saturation | At 28 days
  Using SAFI (SAFI: Index calculated by Oxygen Saturation by Pulse Oximetry / Inspired Fraction of Oxygen)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Red de Salud UC - Christus, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided